CLINICAL TRIAL: NCT00702559
Title: Design the Home Care Platform for the Monitoring of A Hemodialysis Arteriovenous Graft by Intelligent Physiological Signal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: FEMH-96040
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Renal Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Most patients with end-stage renal disease require hemodialysis. An arteriovenous fistula (AVF) or a prosthetic arteriovenous graft (AVG) is the preferred accesses for this. After its surgical creation, the fistular vein immediately faces a tremendous blood flow and the venous lumen is gradually dilated and the wall thickened, producing an access that can be routinely needled and deliver sufficient blood flow for dialysis. However, many hemodialysis patients will experience access stenosis, dysfunction, and even thrombosis, which are the most common complications of a hemodialysis access.

Most physicians, in-charge nurses of the hemodialysis unit, patient, and/or the family use traditional stethoscope as a convenient method to evaluate the patency and function of a hemodialysis access before, during, and after each session of dialysis. The acoustic signal of an access is always affected by environmental noises, non-specific in nature, and the sensitivity to detect stenosis is very low.

With the development and use of electronic stethoscope, the proprietary ambient noise acoustically cancels out an average of 75% of distracting room noise, greatly enhancing overall utility. However, the output acoustic signals are still apprehended by the ear, which is the main source of bias and errors of detection.

Our study purpose is to apply the signal processing technology to transfer the acoustic signals into simple visual signals that provide an easy way to read. It can be used by a professional medical staff, a non-professional person responsible for taking care, or even the patient himself, disability or not, as an early screening detector of stenosis or dysfunction of a hemodialysis access.

ELIGIBILITY:
Inclusion Criteria:

* prosthetic grafts with clinical signs of dysfunctions or malfunctions and were referred for angiographic evaluations.

Exclusion Criteria:

* autologous arteriovenous accesses or known thrombosed accesses.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 50 prosthetic dialysis accesses on upper extremities
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-01

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan